CLINICAL TRIAL: NCT04384211
Title: Smart Bone: An Intelligent Fracture Risk Capture and Management System
Brief Title: QOCA®-Image Medical Platform - Smart VCF Risk Management System
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Quanta Computer Inc. (Unknown)
Responsible Party: Principal Investigator, Wing P Chan, Professor and Chief, Department of Radiology, Wan Fang Hospital, Taipei Medical University, Taipei Medical University WanFang Hospital
Other Study IDs: N201909056
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Compression Fracture
MeSH Terms: conditions — Fractures, Compression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiologists: A computer search of CT scans (2010.01.01-2018.09.30) was performed in Wan Fang Hospital. These CT images were retrospectively reviewed by an experienced radiologist who classified and marked with annotations of vertebral fractures by the Genant's semiquantitative method.
- Smart Bone: The same CT images were separately reviewed and processed by the artificial intelligence system (Smart Bone) by Quanta for compression fractures. The two results, one by the radiologists and the other by artificial intelligence system, will be compared to statistically quantify equivalence (CADe).
  Interventions: Other: Computer Assisted Detection Software For Vertebral Fractures

INTERVENTIONS:
Other: Computer Assisted Detection Software For Vertebral Fractures — A device named Smart Bone that is using CT image retrospectively acquired to entails a second review of CT images with Vertebral Compression Fractures through an interactive AI program developed by Quanta Computer Inc. was applied to the CT images. The device is a computer-aided detection (CADe) software application and is designed to assist radiologists to analyze Spine CT images. The device uses deep learning methods to perform vertebrae detection and classification of images.
  Other Names: Smart Bone
  Groups: Smart Bone

SUMMARY:
This project aims to develop and validate an automatic detection and classification system for vertebral compression fractures on computer tomography (CT) images using an artificial intelligence (AI) system (named Smart Bone) by Quanta.

DETAILED DESCRIPTION:
A computer search of CT scans (2010.01.01-2018.09.30) was performed in Wan Fang Hospital. Those CT images that were retrospectively reviewed by experienced radiologists. The CT scans of 1000-1500 subjects aged 50 and above with and without thoracic or lumbar compression fractures were included in this project for machine learning and deep learning. The control group included those without compression fractures while the patient group were those with compression fractures. Subjects that did not meet the inclusion criteria were excluded.

The cortical layer of the T12-L5 spine images were manually labelled with the labeling software by the the technologists and confirmed the correctness of the image by an experienced radiologist. All the de-linked and completed images were provided to Quanta Computer Inc. for subsequent classification and analysis of AI machines for deep learning to facilitate the development of a system for automatic detection of pressure fractures by CT. This newly developed automatic system will be of valuable clinical impact in assisting radiologists to detect and classify vertebral compression fractures precisely and accurately.

ELIGIBILITY:
Inclusion Criteria:

* Cases with CT examinations acquired between 2010.01-2018.09
* Cases with CT examinations performed with one of the following protocol: whole body, abdomen, and spine
* Cases must be >/= 50 years of age
* Cases with reports from CT examinations ditched as positive or negative compression fractures within a search range from T12 to L5 vertebrae.
* CT images with raw data that are allowed to be reconstructed in axial view with a slice thickness of 1.3 mm
* CT images with raw data that are allowed to be reconstructed in sagittal view with a slice thickness of 2.5 mm

Exclusion Criteria:

* CT images with imaging artifacts, foreign bodies, or implants
* Cases with comorbid conditions, such as infection, cancer metastasis, chronic osteomyelitis, or other nonosteoporotic compression fracture

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 1000-1500 subjects were recruited in both sex, aged 50 and above, and who had come to Wan Fang Hospital for CT scans, including those with or without vertebral compression fractures as the compression fractures group and the control group respectively.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Concordance rate | 2019.06 to 2020.03
  CT Imaging Reporting and Data System descriptors suggested by Smart Bone are in good agreement with those selected by experts. In other words, the CT Imaging Reporting and Data System generated by Smart Bone are not statistically different from the consensus of experts.
  CT Imaging Reporting and Data System Assessment Category Score: The user makes the final decision on the Assessment Category Score. Using this Score, Smart Bone displays the assessment description.
  Grade 0: Normal Vertebrae Grade 1: Mild Fracture, 20-25% Grade 2: Moderate Fracture, 26-40% Grade 3: Severe Fracture, >40%

SECONDARY OUTCOMES:
Accuracy | 2019.06 to 2020.03
  Comparing to the accuracy of CT imaging results by radiologists with and without CADe will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Wing P. Chan, M.D., Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided